CLINICAL TRIAL: NCT02471430
Title: A Phase I-II Pilot Study to Assess the Safety and Efficacy of Combined Administration With Pegylated Interferon-alpha2a and the Histone Deacetylase Inhibitor (HDACi) Panobinostat for Reducing the Residual Reservoir of HIV-1 Infected Cells in cART-Treated HIV-1 Positive Individuals
Brief Title: Reducing the Residual Reservoir of HIV-1 Infected Cells in Patients Receiving Antiretroviral Therapy
Acronym: ACTIVATE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Mathias Lichterfeld, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01 2015P000858; 12049 (Other: Division of AIDS (DAIDS-ES))
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Panobinostat; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Experimental): Participants in Arm A will receive panobinostat as an oral tablet on days 0, 2, and 4 of the treatment week. The dose of panobinostat will be a 15 mg tablet.
  Interventions: Drug: Panobinostat
- Arm B (Experimental): Participants in Arm B will receive one subcutaneous injection of pegylated interferon-alpha2a on day 0. The dose of pegylated IFN-alpha2a will be 180 mcg. Simultaneously with interferon-alpha2a, a 15 mg tablet of panobinostat will be administered on day 0. Participants will also receive panobinostat as an oral tablet on days 2 and 4 of the treatment week.
  Interventions: Drug: Panobinostat; Drug: Pegylated Interferon-alpha2a
- Arm C (Experimental): Participants in Arm C will receive one subcutaneous injection of pegylated interferon-alpha2a on day 0.The dose of pegylated IFN-alpha2a will be 180 mcg.
  Interventions: Drug: Pegylated Interferon-alpha2a

INTERVENTIONS:
Drug: Panobinostat — Panobinostat will be administered orally.
  Other Names: Farydak; LBH589
  Arms: Arm A; Arm B
Drug: Pegylated Interferon-alpha2a — Pegylated Interferon-alpha2a will be administered subcutaneously in one shot.
  Other Names: Pegasys
  Arms: Arm B; Arm C

SUMMARY:
This study is a prospective, open-label, randomized, three-arm, dose-escalation exploratory pilot clinical trial involving HIV-1 infected participants treated with suppressive combination antiretroviral combination therapy (cART). The study will test whether combined treatment with the histone deacetylase inhibitor panobinostat and the immunomodulatory cytokine Interferon-alpha2a can reduce the residual reservoir of HIV-1 infected cells that persist during treatment with currently available antiretroviral drugs.

DETAILED DESCRIPTION:
This study is a prospective, triple-arm, randomized, open-label, dose-escalation exploratory clinical trial involving HIV-1 infected participants treated with suppressive combination antiretroviral combination therapy (cART). The primary objective of this study is to evaluate a new strategy for reducing the residual reservoir of HIV-1 infected cells that persists despite treatment with current HIV drugs. The clinical trial is conducted in the Infectious Diseases Clinical Trials Unit (CTU) at the Massachusetts General Hospital.

The study medication includes two agents: panobinostat is an oral tablet that can reverse HIV-1 latency and awaken HIV from a "sleeping" condition during which it is protected from the human immune system. The second drug is pegylated interferon-alpha2a (IFN-alpha2a), an injectable cytokine that activates the immune system. The combined use of both agents may lead to immune-mediated elimination of HIV-1 infected cells in which viral latency has been reversed by panobinostat.

Participants will be randomized to receive a treatment course with panobinostat alone (Arm A, 4 participants total), panobinostat in combination with pegylated IFN-alpha2a (Arm B, 9 participants total), or pegylated IFN-alpha2a alone (Arm C, 4 participants total). Participants receiving panobinostat will undergo one week of treatment (15mg, dosed every second day on Monday, Wednesday, Friday), followed by three weeks off-treatment. Subcutaneous injections with pegylated IFN-alpha2a will be administered at the start of the week-long treatment course (simultaneously with the first dose of panobinostat for Arm B). ART will be continued during the entire treatment duration in all study participants.

Participants will undergo close monitoring for side effects during the entire time of study participation. The total study duration will be 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide informed consent
* HIV-1 infection prior to entry
* Receiving suppressive ART therapy for a minimum of 24 consecutive months prior to screening with no interruption of therapy (same ART regimen for at least 12 weeks prior to screening)
* Documented suppressed HIV-1 RNA (plasma HIV-1 RNA values <50 copies/ml)
* CD4 T cell count ≥ 400 cells/mm3
* Negative Hepatitis B surface antigen (HBsAg) or Negative HBV DNA PCR
* Negative anti-Hepatitis C virus antibodies (anti-HCV) or negative HCV PCR if anti-HCV antibodies are positive
* Negative TB Test (if positive, completed a recommended treatment course for latent TB)
* Vaccinated for pneumococcal disease within last 5 years
* No clinically significant eye disease
* No evidence of clinical coronary heart disease
* Not pregnant, planning to become pregnant, or breastfeeding
* Willingness to continue to use contraceptives for 90 days after completing treatment
* If male, willingness to use a condom during intercourse while taking panobinostat and total of 80 hours after stopping treatment
* Not pregnant, planning to become pregnant, or breastfeeding
* No evidence of coronary heart disease

Exclusion Criteria:

* HIV-1 RNA > 50 copies/mL within 24 months of screening
* Severe psychiatric disease, chronic liver disease, past or current evidence of immunologically mediated disease
* Severe retinopathy due to diabetes, hypertension, cytomegalovirus or macular degeneration
* Evidence of coronary heart disease
* History of active thyroid disease requiring medication
* Breastfeeding
* Presence of a bacterial, fungal, viral or protozoal infection requiring systemic anti-infective therapy
* Uncontrolled seizure disorders
* History or other evidence of severe illness or other conditions
* History of malignancy of any organ system within the past 5 years
* Female participants who are pregnant or nursing
* History of solid organ transplantation with an existing functional graft
* Use of any immunomodulatory agents within 30 days prior to study enrollment or planned use during the trial
* Active drug or alcohol use or dependence
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the participant in case of participation in the study
* Use of HIV protease inhibitor or other strong or moderately strong CYP3A4 inhibitors
* History of anaphylaxis, allergy or serious adverse reactions to Interferon-alpha2a/Interferon-alpha2b or panobinostat
* Has taken: interleukins, systemic interferons or systemic chemotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Lichterfeld, MD, PhD, Principal Investigator — Massachusetts General Hospital; Daniel R Kuritzkes, MD, Principal Investigator — Massachusetts General Hospital; Rajesh T Gandhi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts, United States

REFERENCES:
- [Background] Rasmussen TA, Tolstrup M, Brinkmann CR, Olesen R, Erikstrup C, Solomon A, Winckelmann A, Palmer S, Dinarello C, Buzon M, Lichterfeld M, Lewin SR, Ostergaard L, Sogaard OS. Panobinostat, a histone deacetylase inhibitor, for latent-virus reactivation in HIV-infected patients on suppressive antiretroviral therapy: a phase 1/2, single group, clinical trial. Lancet HIV. 2014 Oct;1(1):e13-21. doi: 10.1016/S2352-3018(14)70014-1. Epub 2014 Sep 15. PMID 26423811

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 4 | 9 | 4
Completed | 4 | 9 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A (Panobinostat-only Arm): Participants in Arm A will receive panobinostat as an oral tablet on days 0, 2, and 4 of the treatment week. The dose of panobinostat will be a 15 mg tablet.
  Panobinostat: Panobinostat will be administered orally.
- Arm B (Panobinostat + IFNa2a Arm): Participants in Arm B will receive one subcutaneous injection of pegylated interferon-alpha2a on day 0. The dose of pegylated IFN-alpha2a will be 180 mcg. Simultaneously with interferon-alpha2a, a 15 mg tablet of panobinostat will be administered on day 0. Participants will also receive panobinostat as an oral tablet on days 2 and 4 of the treatment week.
  Panobinostat: Panobinostat will be administered orally.
  Pegylated Interferon-alpha2a: Pegylated Interferon-alpha2a will be administered subcutaneously in one shot.
- Arm C (IFN-a2a-only Arm): Participants in Arm C will receive one subcutaneous injection of pegylated interferon-alpha2a on day 0.The dose of pegylated IFN-alpha2a will be 180 mcg.
  Pegylated Interferon-alpha2a: Pegylated Interferon-alpha2a will be administered subcutaneously in one shot.
- Total: Total of all reporting groups
Arm/Group | Arm A (Panobinostat-only Arm) | Arm B (Panobinostat + IFNa2a Arm) | Arm C (IFN-a2a-only Arm) | Total
Number analyzed (Participants) | 4 | 9 | 4 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 9 | 4 | 17
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 49.5 [41 to 60] | 40.4 [26 to 58] | 43.2 [35 to 47] | 43.2 [26 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3
  Male | 3 | 9 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 1 | 8
  Not Hispanic or Latino | 2 | 4 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 3 | 8 | 2 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 9 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Grade ≥ 1 Adverse Events (AEs)
Description: Cumulative frequency and severity of Grade ≥ 1 adverse events, Grade ≥ 1 lab abnormalities or serious adverse events
Time Frame: All adverse events measured from day 1 until day 28 after administration of the first dose of panobinostat and/or interferon-alpha2a was recorded.
Population: all study participants
Measure: Number; unit: events
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 4 | 9 | 4
events | 5 | 26 | 4

2. Primary Outcome: Change in CD4 T Cell-Associated Proviral HIV-1 DNA From Baseline
Description: Operational measurement of CD4 T cells harboring genome-intact HIV-1 DNA, determined by the IPDA assay.
Time Frame: Measured through week 4 after administration of panobinostat and/or interferon-alpha2a
Population: entire study population
Measure: Mean (Standard Error); unit: HIV copies per million CD4 T cells
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 4 | 9 | 4
HIV copies per million CD4 T cells
  baseline | 32.6 (14.1) | 179 (130) | 24 (18.3)
  day 28 | 44.7 (20.2) | 108.4 (79.8) | 18.7 (12.5)

3. Secondary Outcome: Change From Baseline in Histone H3 Acetylation in CD4 T Cells
Description: CD4 T cells expressing acetylated H3, determined by flow cytometry.
Time Frame: measured after last dose of PBT on day 4
Population: entire study cohort
Measure: Mean (Standard Error); unit: Percentage of cells
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 4 | 9 | 4
Percentage of cells
  baseline | 2 (0.64) | 3.1 (0.76) | 5.5 (1.47)
  day 4 | 23.2 (17.15) | 14.7 (3.2) | 8.3 (3.7)

4. Secondary Outcome: Change From Baseline in Levels of CD4 T Cell-associated HIV-1 RNA
Description: total HIV-1 RNA per ug of RNA in CD4 T cells
Time Frame: measured after last dose of PBT on day 4
Population: entire study population
Measure: Mean (Standard Error); unit: HIV RNA copies/ug of RNA
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 4 | 9 | 4
HIV RNA copies/ug of RNA
  baseline | 1055.6 (306.9) | 630.6 (279.3) | 772.5 (302.5)
  day 4 | 1611.2 (596.6) | 1138.4 (583.1) | 958.8 (296)

5. Secondary Outcome: Change From Baseline in Frequency of Activated NKp30+ NK Cells.
Description: the proportion of NK cells expressing NKp30
Time Frame: measured after last dose of PBT on day 4
Population: entire study population
Measure: Mean (Standard Error); unit: percentage of cells
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 4 | 9 | 4
percentage of cells
  baseline | 22.8 (0.9) | 30.9 (3.2) | 21.4 (4.2)
  day 4 | 23 (1.4) | 37.8 (4) | 25.5 (5.6)

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse event definition is as in clinicaltrials.gov
Arm/Group | Arm A | Arm B | Arm C
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/9 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/9 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 9/9 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=4) | Arm B (N=9) | Arm C (N=4)
body aches (General disorders) | 0 (0) | 4 (4) | 1 (1)
fatigue (General disorders) | 0 (0) | 6 (6) | 1 (1)
paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
fever (General disorders) | 0 (0) | 2 (2) | 0 (0)
chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Loose stool (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
increase serum creatinine (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
ECG changes (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT02471430/Prot_SAP_000.pdf